CLINICAL TRIAL: NCT07032766
Title: Assessment of Morbidity and Mortality Following Serratus Anterior Plane Block (SAPB) for Unilateral Rib Fractures
Acronym: SAPB
Status: Recruiting | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-16493
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pain Management; Rib Fracture Multiple; Serratus Anterior Plane Block
Keywords: serratus anterior plane block; rib fractures; mortality; morbidity
MeSH Terms: conditions — Agnosia; Rib Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Serratus Anterior Plane Block (SAPB): Following visualization of the serratus anterior muscle, the latissimus dorsi muscle, and the pleural line, and creating a skin wheel at the puncture site, a 22-gauge 3.5 or 4 inch echogenic PAJUNK® SonoBlock II needle will be inserted just lateral to the transducer at 45 degrees. The needle will be visualized in-plane under real time ultrasound guidance to ensure correct placement between the latissimus dorsi and serratus anterior muscle. 20 ml of bupivacaine hydrochloride 0.25% will be infiltrated into the superficial plane and local anesthetic spread will be observed on ultrasound. Ultrasound images will be obtained pre-procedure, during, and post procedure to demonstrate that the needle tip is away from the pleura and appropriate hydrodissection of muscle fascia occurs.
- Non-SAPB: Patients in this arm will receive IV analgesia, mainly opioid therapy.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of the serratus anterior plane block (SAPB) in adult patients who suffered multiple unilateral anterolateral rib fractures within 24 hours of patient presentation to the emergency department. The main question it aims to answer is:

Does the SAPB for multiple anterolateral rib fractures demonstrate reduction in patient morbidity and mortality, including incidence of pneumonia, length of hospital stay, discharge disposition, and death, as compared to standard analgesic regimens.

The SAPB will be performed if a physician trained in the SAPB is available within 24 hours of injury. If a trained physician is not available and the patient meets inclusion criteria, they will receive parental analgesia with opioid therapy. They will be followed until date of hospital discharge, up until 60 days.

DETAILED DESCRIPTION:
Rib fractures are a common complication of blunt thoracic trauma, reported in 10% of all injured trauma patients. They are associated with significant long-term disability, decreased quality of life, and increased patient morbidity and mortality. Pain from multiple rib fractures can result in reduced respiratory effort, atelectasis, inability to clear secretions, and a reduction in vital capacity. This, in turn, can result in hypoxemia, pneumonia, and acute respiratory failure. Adequate and early pain management is therefore crucial to provide symptomatic relief, decrease splinting, and prevent secondary respiratory complications.

While systemic analgesia, notably opioids, are frequently used in the emergency department (ED) for pain control, they are associated with poor side effect profiles. Opioids place patients at risk for delirium, chronic addiction, respiratory depression, and constipation. Traditional regional anesthesia techniques, including paravertebral, intercostal and epidural injections, are resource-intensive, time consuming, limited in dermatomal distribution and associated with significant potential complications (diaphragmatic complications, local anesthetic toxicity, vasovagal syncope, pneumothoraces). Such techniques are not feasible in the ED. Ultrasound-guided fascial plane blocks have thus emerged as an alternative tool for proper pain control in patients with rib fractures in the ED. Fascial plane blocks include the serratus anterior plane block (SAPB) and the erector spinae plane block (ESPB).

The SAPB has demonstrated efficacy in providing safe analgesia for anterolateral rib fractures, while the ESPB has demonstrated efficacy in pain relief of posterior rib fractures. A benefit of SAPB is that it can be performed in the supine position, in contrast to other regional anesthesia techniques. The SAPB utilizes a linear transducer to identify the serratus anterior muscle and instill local anesthetic into the fascial plane overlying the muscle. The anesthetic targets the lateral cutaneous branches of the intercostal nerves, with a wide distribution centered around T3-T8. The anesthetic may also block the long thoracic and thoracodorsal nerve if injected superficial to the serratus anterior muscle. Recent studies have demonstrated improvement in chest wall pain scores and incentive spirometry (IS) following SAPB in adult patients with rib fractures. No SAPB attributed complications have been reported, likely related to the clear landmarks of the procedure and injection of anesthetic into a compartment distant from major vasculature. To date, no studies have investigated the effects of SAPB on morbidity and mortality as compared to standard oral or intravenous (IV) analgesics in patients with multiple rib fractures. The authors aim to prospectively assess whether SAPB for multiple anterolateral rib fractures demonstrates reduction in key outcome measures as compared to standard analgesic regimens. The study is a prospective cohort study which will take place at a single urban level 1 trauma center.

For patients who meet inclusion and exclusion criteria, SAPB will be utilized as part of a multimodal analgesia strategy if an emergency physician trained in the procedure is present in the ED within 24 hours of injury. If a SAPB-trained emergency physician is not available, the patient will be placed in the non-SAPB group. Patients will be enrolled in the study by clinicians participating in their care who are involved in performance of the SAPB. Morbidity and mortality, the composite outcome measures, will be assessed through various primary outcome measures, each indexed separately (see Outcome Measures section).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age being treated in the Emergency Department at Jacobi Medical Center
* Presenting within 24 hours of injury
* Patient with 2 or more unilateral, anterior or lateral rib fractures
* Able to provide consent (patient or health care proxy)
* Clinical team believes the patient will require inpatient admission at the time of enrollment

Exclusion Criteria:

* Patients in traumatic arrest or hemodynamic instability
* Patient expected to be discharged from the hospital within 24 hours
* Prisoner
* Pregnancy
* Children less than 18 years of age
* The patient is known or is suspected to be allergic to anesthetic
* Significant pain from another traumatic and distracting injury
* Patients without the ability to consent (or no health care proxy to consent)
* Patients with bilateral or posterior rib fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include a cohort of patients presenting within 24 hours of injury with two or more unilateral, anterior or lateral rib fractures requiring opioid analgesia that would be admitted to the trauma service at a single urban level 1 trauma center. The authors anticipate recruitment of 200 participants over the course of a study duration of 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Hospital Acquired Pneumonia (HAP) Events | From time of ED arrival until hospital discharge, up until 90 days
  The number of patients of hospital acquired pneumonia events will be summarized by study arm/group using basic descriptive statistics.
Days of Hospital Length of Stay | ED arrival to hospital discharge, up until 90 days
  For purposes of this study, length of hospital stay will be defined as the total duration of admission and will be recorded in total number of days (from ED admission to discharge) and summarized by study arm/group using basic descriptive statistics. Discharge may include to acute rehabilitation (located in the hospital but not considered in calculation for length of stay).
Discharge Disposition | ED admission to discharge , up until 90 days
  Discharge Disposition will encompass the location to which the patient is discharged (i.e., home, home with Physical Therapy (PT), subacute rehabilitation, acute rehabilitation, or deceased). Disposition types will be categorically itemized and summarized by study arm/group.
Length of stay (Days) in the Intensive Care Unit (ICU) | ED admission to hospital discharge, up until 90 days
  For purposes of this study, ICU length of stay will be defined as the total number of days of admission to an ICU and will be summarized by study arm/group using basic descriptive statistics. If a patient is discharged from the ICU and subsequently returns to the ICU, the total duration of admission will be aggregated.
Cause of death | ED admission until hospital discharge, up until 90 days
  If a patient is "discharged as deceased" (see prior outcome measure) the cause of death will be recorded, if known, and summarized by study arm/group.

SECONDARY OUTCOMES:
Pain Intensity | Baseline (initial evaluation) and 30 and 60 minutes after SAPB is performed
  Patient-reported pain scores will be recorded using an 11-point Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain) such that higher scores are associated with increased pain intensity. Pain scores will be recorded upon initial evaluation (baseline) and 30 and 60 minutes following SAPB. Scores will be summarized by study arm/group using basic descriptive statistics.
Number of patients per group that required additional analgesia | Up until 24 hours after the initial block or IV opioid medication administration
  The number of patients that required additional opioid analgesia after the administration of IV opioid medications or initial (SAPB) block will be assessed and summarized by study arm/group using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Montenegro, MD, Principal Investigator — Albert Einstein College of Medicine, Jacobi medical center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, Statistical Analysis Plan (SAP), and Informed Consent Form (ICF) will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 10 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Lin J, Hoffman T, Badashova K, Motov S, Haines L. Serratus Anterior Plane Block in the Emergency Department: A Case Series. Clin Pract Cases Emerg Med. 2020 Jan 21;4(1):21-25. doi: 10.5811/cpcem.2019.11.44946. eCollection 2020 Feb. PMID 32064417
- [Background] Schnekenburger M, Mathew J, Fitzgerald M, Hendel S, Sekandarzad MW, Mitra B. Regional anaesthesia for rib fractures: A pilot study of serratus anterior plane block. Emerg Med Australas. 2021 Oct;33(5):788-793. doi: 10.1111/1742-6723.13724. Epub 2021 Jan 29. PMID 33511786
- [Background] Serra S, Santonastaso DP, Romano G, Riccardi A, Nigra SG, Russo E, Angelini M, Agnoletti V, Guarino M, Cimmino CS, Spampinato MD, Francesconi R, Iaco F. Efficacy and safety of the serratus anterior plane block (SAP block) for pain management in patients with multiple rib fractures in the emergency department: a retrospective study. Eur J Trauma Emerg Surg. 2024 Dec;50(6):3177-3188. doi: 10.1007/s00068-024-02597-6. Epub 2024 Jul 17. PMID 39020130
- [Background] Paul S, Bhoi SK, Sinha TP, Kumar G. Ultrasound-Guided Serratus Anterior Plane Block for Rib Fracture-Associated Pain Management in Emergency Department. J Emerg Trauma Shock. 2020 Jul-Sep;13(3):208-212. doi: 10.4103/JETS.JETS_155_19. Epub 2020 Sep 18. PMID 33304071
- [Background] Hernandez N, de Haan J, Clendeninn D, Meyer DE, Ghebremichael S, Artime C, Williams G, Eltzschig H, Sen S. Impact of serratus plane block on pain scores and incentive spirometry volumes after chest trauma. Local Reg Anesth. 2019 Aug 2;12:59-66. doi: 10.2147/LRA.S207791. eCollection 2019. PMID 31447581
- [Background] Kring RM, Mackenzie DC, Wilson CN, Rappold JF, Strout TD, Croft PE. Ultrasound-Guided Serratus Anterior Plane Block (SAPB) Improves Pain Control in Patients With Rib Fractures. J Ultrasound Med. 2022 Nov;41(11):2695-2701. doi: 10.1002/jum.15953. Epub 2022 Feb 2. PMID 35106815
- [Background] Kumar G, Kumar Bhoi S, Sinha TP, Paul S. Erector spinae plane block for multiple rib fracture done by an Emergency Physician: A case series. Australas J Ultrasound Med. 2020 Aug 30;24(1):58-62. doi: 10.1002/ajum.12225. eCollection 2021 Feb. PMID 34760612
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Picard J, Meek T. Complications of regional anaesthesia. Anaesthesia. 2010 Apr;65 Suppl 1:105-15. doi: 10.1111/j.1365-2044.2009.06205.x. PMID 20377552
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Sadauskas V, Fofana M, Brunson D, Choi J, Spain D, Quinn JV, Duanmu Y. Serratus anterior plane block improves pain and incentive spirometry volumes in trauma patients with multiple rib fractures: a prospective cohort study. Trauma Surg Acute Care Open. 2024 Jun 13;9(1):e001183. doi: 10.1136/tsaco-2023-001183. eCollection 2024. PMID 38881827
- [Background] Choi J, Khan S, Hakes NA, Carlos G, Seltzer R, Jaramillo JD, Spain DA. Prospective study of short-term quality-of-life after traumatic rib fractures. J Trauma Acute Care Surg. 2021 Jan 1;90(1):73-78. doi: 10.1097/TA.0000000000002917. PMID 32925583
- [Background] Choi J, Khan S, Sheira D, Hakes NA, Aboukhater L, Spain DA. Prospective study of long-term quality-of-life after rib fractures. Surgery. 2022 Jul;172(1):404-409. doi: 10.1016/j.surg.2021.11.026. Epub 2021 Dec 27. PMID 34969527
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614